CLINICAL TRIAL: NCT01755819
Title: Clinical Outcome and Tunnel Widening After Hamstring Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Computed Tomography - Based Trial Comparing Aperture With Cortical Fixation
Brief Title: Outcome and Tunnel Widening After ACL Reconstruction: Comparison of Aperture and Cortical Fixation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Dr. René El Attal, Principal Investigator, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACL Tightrope vs. Biocomposite
Record Dates: First submitted 2012-12-04; First posted 2012-12-24 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: ACL Anterior Cruciate Ligament Injury; Outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biocomposite interference screw (Other): Thirty patients treated with ACL reconstruction and graft fixation is performed using Biocomposite interference screw on tibial and femoral side. Patients are randomized to one of the two study arms.
  Interventions: Device: Biocomposite interference screw
- Extracortical ACL Tightrope fixation (Other): Thirty patients treated with ACL reconstruction and graft fixation is performed using extracortical ACL Tightrope fixation on tibial and femoral side. Patients are randomized to one of the two study arms.
  Interventions: Device: Extracortical ACL Tightrope fixation

INTERVENTIONS:
Device: Biocomposite interference screw
  Arms: Biocomposite interference screw
Device: Extracortical ACL Tightrope fixation
  Arms: Extracortical ACL Tightrope fixation

SUMMARY:
Background:

Failure of graft incorporation and tunnel widening (TW) after anterior cruciate ligament (ACL) reconstruction has been frequently reported in the literature. The etiology of TW is still not fully understood.

Patients and Methods:

This is a prospective randomized study including 60 patients, conducted in a Level I trauma center in Innsbruck, Austria. The study protocol was approved by the hospital ethics committee. This study is planned and conducted following the Consolidated Standards on Reporting Trials (CONSORT) guidelines. Aperture fixation is performed using BioComposite interference screws (Arthrex, Naples, FL). Extracortical fixation is performed using the ACL Tightrope (Arthrex, Naples, FL). TW is measured on CT scan postoperative, after 6 and 24 months. Clinical outcome is determined at 1, 2 after reconstruction, IKDC with KOOS Knee-related QoL subscale, Lysholm, Tegner Activity scores, hop tests and KT-1000 measurements are performed.

Hypothesis:

The purpose of this randomized controlled trail is to determine the influence of two different fixation methods on TW and clinical outcome after anatomic ACL reconstruction using hamstring graft in young and active patients.

DETAILED DESCRIPTION:
The study is a randomized controlled clinical trial and will be conducted at the Traumasurgery Innsbruck. Two different surgical methods are tested: ACL Tightrope reconstruction VS Biocomposite interference screws.

Following eligibility criteria have to be met:

1. Age 18 -40 years
2. ACL insufficiency diagnosed by clinical examination (positive Lachman test and/or pivot shift test) and MRI (complete tear)
3. Not more than 12 month after trauma to the knee
4. Tegner Score 5 to 10

Not eligible if:

1. Earlier major knee injury to the index knee
2. Previous knee surgery (except diagnostic arthroscopy) to index knee
3. Associated knee fractures
4. Associated PCL injury, complete MCL or LCL tear
5. Concomitant severe injury to contra-lateral knee at time of assessment
6. Injury to the lateral/posterolateral ligament complex with increased laxity (positive dial test and external rotation thigh foot angle test),
7. Pregnancy and scope to become within next time
8. A history of deep vein thrombosis (DVT) or a disorder of the coagulative system
9. Claustrophobia
10. General systemic disease affecting physical function, any other condition or treatment interfering with the completion of the trial, including patients with metal devices, pacemaker or motion disorders
11. Chronic systemic use of steroids

Following inclusion and exclusion criteria have to be met:

Inclusion:

1. The ACL injury can be either "isolated" or combined with one or several of the following injuries visualized on MRI and/or arthroscopy:

   * A meniscus tear that is either left untreated or treated with a partial resection
   * A small, stable meniscus tear treated with fixation, but fixation not interfering with the rehabilitation protocol
   * Cartilage changes verified on MRI with arthroscopically determine intact surface
2. A radiographic examination with normal joint status or combined with either one of the following finding:

   * A small avulsed fragment located laterally, usually described as a Second fracture
   * JSN grade 1 or osteophytes grade 1 as determined by the OARSI atlas (Altman et al. 1995)
3. Agreement to participate in the study and signed informed consent prior to inclusion.

Exclusion:

1.Presence of one of the following associated injuries to the index knee as visualized on MRI and/or arthroscopy:

* An unstable longitudinal meniscus tear that requires repair and where the following postoperative treatment (i.e. bracing and limited ROM) interferes with the rehabilitation protocol
* Bi-compartmental extensive meniscus resection
* A cartilage injury representing a full thickness loss down to bone
* A total rupture of MCL/LCL as visualized on MRI

A power analysis was performed, estimating that a minimum of 34 patients (17 in each group) would be required to obtain a power more than 80%.

ELIGIBILITY:
Inclusion Criteria:

1. The ACL injury can be either "isolated" or combined with one or several of the following injuries visualized on MRI and/or arthroscopy:

   * A meniscus tear that is either left untreated or treated with a partial resection
   * A small, stable meniscus tear treated with fixation, but fixation not interfering with the rehabilitation protocol
   * Cartilage changes verified on MRI with arthroscopically determine intact surface
2. A radiographic examination with normal joint status or combined with either one of the following finding:

   * A small avulsed fragment located laterally, usually described as a Second fracture
   * JSN grade 1 or osteophytes grade 1 as determined by the OARSI atlas (Altman et al. 1995)
3. Agreement to participate in the study and signed informed consent prior to inclusion.

Exclusion Criteria:

1.Presence of one of the following associated injuries to the index knee as visualized on MRI and/or arthroscopy:

* An unstable longitudinal meniscus tear that requires repair and where the following postoperative treatment (i.e. bracing and limited ROM) interferes with the rehabilitation protocol
* Bi-compartmental extensive meniscus resection
* A cartilage injury representing a full thickness loss down to bone
* A total rupture of MCL/LCL as visualized on MRI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change of tunnel volume and diameter from baseline up to 2 year follow up | 1-2 days before (knee) operation, 6 months FU, 2 year FU
  CT tunnel measurements are conducted. Tunnel volume are calculated by CT volumetry measured in mm³ and tunnel diameter is measured in mm.

SECONDARY OUTCOMES:
Clinical outcome: international knee score evaluating objective and subjective knee outcome variables | 1-2 days before (knee)operation, 6 months FU, 1 year FU, 2 year FU
  Clinical outcome measured by IKDC (INTERNATIONAL KNEE DOCUMENTATION COMMITTEE) Subjective questionnaire (symptoms, sports activity, knee function): scaled from 0-100.
  Objective evaluation form (radiological assessment of cartilage and menisci, functional knee examination, range of motion): scaled A-D
Clinical outcome: influence on quality of life after knee ACL reconstruction | 1-2 days before (knee)operation, 6 month FU, 1 year FU, 2year FU
  Clinical outcome measured by KOOS Knee related QoL subscale
Clinical outcome: subjective evaluation of knee function | 1-2 days before (knee)operation, 6 months FU, 1 year FU, 2 year FU
  Clinical outcome measured by Lysholm Score: subjective questionnaire
Clinical outcome: return to sports activity | 1-2 days before (knee)operation, 6 months FU, 1 year FU, 2 year FU
  Clinical outcome measured by Tegner Activity scores: sports activity level
Clinical outcome: strength in single leg jumping after ACL reconstruction | 1-2 days before (knee)operation, 6 months FU, 1 year FU, 2 year FU
  Single leg hop test measured in cm. Comparing the injured and healthy knee.
Clinical outcome: objective knee anterior stability | 1-2 days before (knee)operation, 6 months FU, 1 year FU, 2 year FU
  Clinical outcome measured by KT1000 arthrometer measurements in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Rene El Attal, Dr., Principal Investigator — Medical University Innsbruck (Traumasurgery)
Locations (1):
- Medical University Innsbruck (Traumasurgery), Innsbruck, Tyrol, Austria

REFERENCES:
- [Derived] Eichinger M, Ploner M, Degenhart G, Rudisch A, Smekal V, Attal R, Mayr R. Tunnel widening after ACL reconstruction with different fixation techniques: aperture fixation with biodegradable interference screws versus all-inside technique with suspensory cortical buttons. 5-year data from a prospective randomized trial. Arch Orthop Trauma Surg. 2023 Nov;143(11):6707-6718. doi: 10.1007/s00402-023-05001-x. Epub 2023 Aug 5. PMID 37542556
- [Derived] Mayr R, Smekal V, Koidl C, Coppola C, Eichinger M, Rudisch A, Kranewitter C, Attal R. ACL reconstruction with adjustable-length loop cortical button fixation results in less tibial tunnel widening compared with interference screw fixation. Knee Surg Sports Traumatol Arthrosc. 2020 Apr;28(4):1036-1044. doi: 10.1007/s00167-019-05642-9. Epub 2019 Aug 1. PMID 31372680